CLINICAL TRIAL: NCT01251094
Title: Dementia Registry for Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DRM99-IRB-233
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Dementia; Parkinson's Disease
Keywords: Dementia; Parkinson's; impairment; Dementia Registry for Parkinson's Disease
MeSH Terms: conditions — Dementia; Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Background

Cognitive impairment in Parkinson's disease (PD) is common, even in the early stage of this disease.The cumulative prevalence of dementia associated with Parkinson's disease (PDD) is as high as 80% in a recent 8-year prospective study. However, some kinds of cognitive impairment are not apparent and the value of self-report cognitive decline became limited. In other words, some cognitive impairment may be detected by cognitive tests rather than self-report of the symptoms.The early intervention of the cognitive impairment may be helpful for these patients. Neuropsychiatric symptoms(NPSs) are also common in PD and PDD patients. The severity of NPSs contributes to reduced quality of life and distress for caregivers. Previous studies showed some different clinical phenotypes of NPSs in PD or PDD patients. Among the NPSs, hallucination was considered a critical factor of cognitive dysfunction in PD and PDD patients. The co-occurrence of NPSs in PD and PDD patients has limited evidence now.

Purpose

To establish the screening tools for early detecting the PD patient with cognitive impairment; exam the diagnostic value of MoCA and other cognitive tests in PD with mild cognitive impairment, possible PDD, and probable PDD; understand neuropsychiatric symptoms (NPSs) in these different patient groups; exam the relationship between each NPS and each domain of cognitive dysfunction.

Methods

In order to exam the cognitive dysfunction in PDD (attention, executive function, visuo-spatial function, and memory), several tests are performed. A 32-item cognitive decline questionnaire will be used to screen the cognitive impairment in subjects. Mini-Mental state examination (MMSE) and Montreal cognitive assessment (MoCA)are used for cognitive evaluation. The detail evaluation of each domain is specified asfollowing: (1) Attention (WAIS-R digit span), (2) Memory (12-item word recall test),(3) Executive function (category verbal fluency), (4) Visuospatial function (cube copying and clock drawing). The motor symptoms severity of the PD will be evaluated by the Hoehn & Yahr stage and motor portion of the Unified Parkinson's Disease Rating Scale (UPDRS). The neuropsychiatric symptoms will be recorded by Neuropsychiatric Inventory Questionnaire (NPI-Q). The daily living activity will beevaluated by modified Lawton's instrumental activities of daily living scale (IADL)and pill questionnaire. Subjects also receive 15-item Geriatric Depression Scale(GDS-S) to evaluate the mood status. The clinician's diagnosis of dementia will be based on the diagnostic criteria of DSM-IV, which will be compared with the PDDdiagnostic criteria proposed by MDS in 2007. The investigators will also try to develop a PDDscreening questionnaire.

Expected results

Cognitive impairment and dementia of PD patients will be ascertained by the cognitive test battery. The screening questionnaire will be established. The heterogeneity of NPSs in PD and PDD will be evaluated. The PDD screening questionnaire will help the clinician to diagnose the patients.

ELIGIBILITY:
Inclusion Criteria:

1. The patient who is diagnosed as clinical PD with and without dementia according to the DSM-IV criteria [3] will be invited for this study. The diagnosis of clinical PD is according to the UK Parkinson's Disease Society Brain Bank clinical diagnostic criteria [17]. The initial symptom more than one year of clinical PD will be invited for this study.
2. A reliable caregiver who lives with the subjects or has at least 10 hours/week of contact with the subject.
3. Males and females between the ages of 50 and 90 years, inclusive.
4. Adequate visual and auditory abilities to perform all aspects of the study assessments.

Exclusion Criteria:

Presence of any of the following criteria will exclude the subject from enrollment in the study:

1. Significant neurological disease other than PD that may affect cognition.
2. Current clinically important systemic illness that is likely to result in deterioration of the subject's condition or affect the subject's safety during the study.
3. History of clinically evident stroke.
4. History of seizures within the past 5 years
5. Myocardial infarction within the past one year prior to screening
6. Current DSM-IV-TR diagnosis of substance abuse or dependence (including alcohol abuse or dependence but excluding nicotine dependence) or history of substance dependence within the past 2 years to screening.
7. Regular use of anticholingeric drugs within 60 days prior to screening.
8. The subject received deep brain stimulation

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's Disease patients.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, North Area, Taiwan